CLINICAL TRIAL: NCT04308902
Title: OptiMoM Grows Up: 5.5-year Follow-up of the OptiMoM Fortifier Study
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Sinai Health System (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Deborah O'Connor, Senior Associate Scientist, The Hospital for Sick Children
Other Study IDs: 1000065339
Record Dates: First submitted 2020-03-11; First posted 2020-03-16 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Infant, Very Low Birth Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children previously enrolled in the OptiMoM Fortifier Study: This is an observational study of children who were previously enrolled in a trial (Bovine vs. Human Milk-Based Fortifier Study) between 2014 and 2016 during which time they were randomized to have their feeds (mother's own milk or pasteurized donor breastmilk) nutrient enriched with a human milk-based fortifier or a bovine protein-based fortifier.
  Interventions: Other: VLBW
- Term-born Comparison: This is an observational study of children born at full term (>= 37 weeks gestation) and weighing more than 2500g. These children will be recruited from the communities in which the OptiMoM participants live.
  Interventions: Other: Term-born Comparison

INTERVENTIONS:
Other: VLBW — Participants previously enrolled in the Bovine vs. Human Milk-Based Fortifier Study
  Groups: Children previously enrolled in the OptiMoM Fortifier Study
Other: Term-born Comparison — Children born >=37 weeks gestation and weighing more than 2500g
  Groups: Term-born Comparison

SUMMARY:
In Canada, the leading cause of long-term disability in children is being born at very low birth weight (VLBW). To help improve outcomes, nutrition is a modifiable aspect of infant care. Mother's milk is the optimal way to feed VLBW infants; however, many need a supplement of donor milk or preterm formula as not enough mother's milk is available. As the ideal supplement for prolonged feeding and its long-term effects is currently unknown, this study is a prospective follow-up of infants born VLBW who were fed mother's own milk or pasteurized donor breastmilk nutrient enriched with a human milk-based fortifier or a bovine protein-based fortifier. Intakes of donor milk, fortifier type, macronutrients and fatty acids will be explored. Areas of development to be assessed include: cognition, language, motor skills, and body composition. This study will also cross-sectionally examine aspects of eating behaviours, food parenting and the home environment (e.g., stress, home chaos, family functioning) with a term-born comparison. A DNA biorepository will also be created.

ELIGIBILITY:
Inclusion Criteria:

* Children who were enrolled in the Bovine vs. Human Milk-Based Fortifier Study (NCT02137473)
* Children who were born >=37 weeks gestation and weighing > 2500g [Term-born comparison group]

Exclusion Criteria:

* For term-born comparison only: a child with any chromosomal or congenital anomaly affecting growth

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Very low birth weight infants previously enrolled in the Bovine vs. Human Milk-Based Fortifier Study (NCT02137473) and a comparison group of children born full-term (>=37 weeks gestation) and weighing >2500g.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Full-Scale Intelligence Quotient (IQ) | 5.5 years of age
  Measured using the assessor-administered Wechsler Preschool and Primary Scale of Intelligence-IV (WPPSI-IV). The WPPSI-IV Full-scale IQ and all composite sub-scales are standardized to a mean of 100, with a standard deviation of 15. Higher scores indicate superior performance.
Growth | 5.5 years of age
  Growth as assessed by weight in kilograms (kg) and height in meters (m) measured by trained staff to assess body mass index (BMI). BMI will be the ratio of weight (kg) to the square of height (m).

SECONDARY OUTCOMES:
Verbal Comprehension Index | 5.5 years of age
  Measured using the assessor-administered Wechsler Preschool and Primary Scale of Intelligence-IV (WPPSI-IV). The WPPSI-IV composite sub-scales are standardized to a mean of 100, with a standard deviation of 15. Higher scores indicate superior performance.
Visual Spatial Index | 5.5 years of age
  Measured using the assessor-administered Wechsler Preschool and Primary Scale of Intelligence-IV (WPPSI-IV). The WPPSI-IV composite sub-scales are standardized to a mean of 100, with a standard deviation of 15. Higher scores indicate superior performance.
Working Memory Index | 5.5 years of age
  Measured using the assessor-administered Wechsler Preschool and Primary Scale of Intelligence-IV (WPPSI-IV). The WPPSI-IV composite sub-scales are standardized to a mean of 100, with a standard deviation of 15. Higher scores indicate superior performance.
Fluid Reasoning Index | 5.5 years of age
  Measured using the assessor-administered Wechsler Preschool and Primary Scale of Intelligence-IV (WPPSI-IV). The WPPSI-IV composite sub-scales are standardized to a mean of 100, with a standard deviation of 15. Higher scores indicate superior performance.
Vocabulary Acquisition Index | 5.5 years of age
  Measured using the assessor-administered Wechsler Preschool and Primary Scale of Intelligence-IV (WPPSI-IV). The WPPSI-IV composite sub-scales are standardized to a mean of 100, with a standard deviation of 15. Higher scores indicate superior performance.
Processing Speed Index | 5.5 years of age
  Measured using the assessor-administered Wechsler Preschool and Primary Scale of Intelligence-IV (WPPSI-IV). The WPPSI-IV composite sub-scales are standardized to a mean of 100, with a standard deviation of 15. Higher scores indicate superior performance.
Body Composition | 5.5 years of age
  Trained staff will measure body composition (e.g., % fat mass, % fat-free mass) using air displacement plethysmography, i.e., BODPOD™.
Body Composition | 5.5 years of age
  Trained staff will measure body composition using bicep, tricep, subscapular and superilliac skinfold thicknesses.
Diet Quality | 5.5 years of age
  Diet Quality as measured using the Healthy Eating Index calculated from two 24-hour recalls conducted by trained staff. Scores on the Healthy Eating Index range from 0-100 with higher scores indicated higher diet quality.
Waist circumference | 5.5 years of age
  Trained staff will measure waist circumference (cm) at the midpoint between the top of the iliac crest and lowest rib.
Blood pressure | 5.5 years of age
  Trained staff will measure blood pressure using an automated sphygmomanometer.

OTHER OUTCOMES:
Affect Recognition domain | 5.5 years of age
  Measured using the assessor-administered Developmental Neuropsychological Assessment-Second Edition (NEPSY-II). Scaled scores for each subtest consist of a mean of 10 and a standard deviation of 3 (range of 1-19). Higher scores indicate superior performance.
Inhibition domain | 5.5 years of age
  Measured using the assessor-administered Developmental Neuropsychological Assessment-Second Edition (NEPSY-II). Scaled scores for each subtest consist of a mean of 10 and a standard deviation of 3 (range of 1-19). Higher scores indicate superior performance.
Design Fluency domain | 5.5 years of age
  Measured using the assessor-administered Developmental Neuropsychological Assessment-Second Edition (NEPSY-II). Scaled scores for each subtest consist of a mean of 10 and a standard deviation of 3 (range of 1-19). Higher scores indicate superior performance.
Statue domain | 5.5 years of age
  Measured using the assessor-administered Developmental Neuropsychological Assessment-Second Edition (NEPSY-II). Scaled scores for each subtest consist of a mean of 10 and a standard deviation of 3 (range of 1-19). Higher scores indicate superior performance.
Visual-Motor Integration | 5.5 years of age
  Measured using the assessor-administered Beery-Buktenica Developmental Test of Visual-Motor Integration (Beery VMI). Standard scores with a mean of 100 and a standard deviation of 15 will be reported. Higher scores on the Beery VMI indicate superior performance.
Social-Emotional Functioning | 5.5 years of age
  Social-Emotional functioning as measured by parent-report using the Social Responsiveness Scale Second Edition (SRS-2). T-scores on the SRS-2 have a mean of 50 and standard deviation of 10. Higher scores are associated with more severe social impairments.
Behaviour and Emotional Response | 5.5 years of age
  Behaviour and Emotional Response as measured by parent-report using the Behavior Assessment System for Children-Third Edition (BASC-3). Scores are expressed as T-scores with a mean of 50 and standard deviation of 10. Higher values indicate increased risk for composites of clinical scales and lower risk for the composite of adaptive scales.
Executive Functioning | 5.5 years of age
  Executive Functioning as measured by parent-report using the Behavioral Rating Inventory of Executive Function (BRIEF). T-scores have a mean of 50 and a standard deviation of 10. Higher scores indicate a potential problematic area of clinical significance.
Sensory Processing | 5.5 years of age
  Sensory Processing related to auditory, visual, touch, movement, body position and oral processing as measured by parent-report using the Sensory Profile Second Edition (Sensory Profile-2). Higher scores indicating higher sensitivity in each category.
Gross Motor Development | 5.5 years of age
  Measured using the assessor-administered Movement Assessment Battery for Children Second Edition (Movement ABC-2). Higher scores indicate superior performance.
Influence of the diet on epigenetic changes | 5.5 years of age
  Assessed using a buccal cell biorepository.
Influence of genetics on taste | 5.5 years of age
  Assessed using a buccal cell biorepository.
Fatty acid status | 5.5 years of age
  Assessed using a buccal cell biorepository.
Children's eating behaviours and dietary intake | 5.5 years of age
  Assessed using direct observation during a standardized lunch protocol.
Children's eating behaviours | 5.5 years of age
  Assessed by parent-report using the Child Eating Behaviour Questionnaire (CEBQ). The CEBQ is made up of eight scales: Food responsiveness, Emotional over-eating, Enjoyment of food, Desire to drink, Satiety responsiveness, Slowness in eating, Emotional under-eating, and Food fussiness. Higher scores indicate higher frequency behaviour.
Food parenting and parent dietary intake | 5.5 years of age
  Assessed using direct observation during a standardized lunch protocol.
Food parenting | 5.5 years of age
  Assessed by parent-report using the Comprehensive Feeding Practices Questionnaire (CFPQ). The questionnaire contains 12 scales: 'Encourage Balance and Variety', 'Environment', 'Involvement', 'Modeling', 'Monitoring', 'Teaching about Nutrition', 'Emotion Regulation', 'Food as Reward', 'Pressure', 'Child Control', 'Restriction for Health' and 'Restriction for Weight Control'; higher scores indicate higher frequency behaviour.
Composition and community structure of the gastrointestinal microbiota | 5.5 years of age
  High-throughput sequencing of microbial DNA from stool samples
Parent and child stress | 5.5 years of age
  Measured using cortisol levels obtained from hair samples collected from both parent and child at the posterior vertex.
Parental stress | 5.5 years of age
  Measured by parent-report using the Parent Distress sub-scale of the Parenting Stress Index Short Form (PSI-SF). Higher scores indicate higher levels of parental distress.
Home environment- Family Functioning | 5.5 years of age
  Family functioning will be measured by parent-report using the General Functioning sub-scale of the Family Assessment Device (FAD). Higher scores indicate lower levels of functioning (problem solving, communication, etc.).
Home environment- Home Chaos | 5.5 years of age
  Home Chaos will be measured by parent-report using the Confusion, Hubbub and Order Scale (CHAOS). Higher scores indicate a more chaotic home environment.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Walton K, Hopperton KE, Lambis A, Law N, Vaz S, Kiss A, Unger SL, O'Connor DL. Caregiver feeding practices, dietary intake and weight status of very low birthweight infants compared to term-born peers at school-entry. Appetite. 2026 Feb 1;217:108338. doi: 10.1016/j.appet.2025.108338. Epub 2025 Oct 8. PMID 41072552